CLINICAL TRIAL: NCT06961071
Title: Parathyroid Allotransplant for Treatment of Hypoparathyroidism: PATTH
Brief Title: Parathyroid Allotransplant for Treatment of Hypoparathyroidism
Acronym: PATTH
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter Stock (Other)
Responsible Party: Sponsor-Investigator, Peter Stock, Professor of Surgery (MD, PhD), University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-40309
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hypoparathyroidism; Hypoparathyroidism Postprocedural; Hypoparathyroidism Post-surgical
Keywords: hypoparathyroidism; parathyroid hormone; PTH; serum calcium; phosphorus
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parathyroid Allotransplant (Experimental): Parathyroid Allotransplant to treat hypoparathyroidism
  Interventions: Biological: Parathyroid Allotransplant

INTERVENTIONS:
Biological: Parathyroid Allotransplant — Parathyroid Allotransplant

SUMMARY:
This study is being done to see if transplanting parathyroid tissue into the forearm will help hypo-parathyroid patients achieve parathyroid hormone (PTH) levels that would help normalize their serum calcium and phosphorus levels. The parathyroid tissue used in this study will come from cadaveric tissues that were donated at the time of the death of the donor(s).

DETAILED DESCRIPTION:
The company that makes the parathyroid hormone NATPARA will no longer be making the product by the end of 2024 which is one of the reasons the investigators are doing this study: to see if parathyroid transplantation is another way to treat hypoparathyroidism. This procedure is investigational and one of the first times the procedure is being done in humans. It is not approved by the FDA.

ELIGIBILITY:
Inclusion Criteria Only subjects who meet all of the following criteria are eligible for enrollment.

1. Subjects age 18 or older.
2. Subjects who are able to provide written informed consent and to comply with study procedures.
3. Clinical history and laboratory data compatible with hypoparathyroidism (HypoPT) as defined by hypocalcemia and documented PTH levels below the normal range on two occasions greater than 2 weeks apart and 12 months after surgery, requiring large doses of activated vitamin D and oral calcium (>1G) daily, or currently on PTH (1-84) injections and with ongoing symptomatology due to hypocalcemia and variable degree of biochemical control
4. No history of immunodeficiency (e.g., opportunistic infections) that could be exacerbated by immunosuppression.
5. Up to date immunizations per the University of California, San Francisco (UCSF) standard of care for organ transplantation, including influenza, pneumococcal, hepatitis B, and tetanus-diptheria

Exclusion Criteria Subjects who meet any of the following criteria are not eligible for enrollment

1. Presence of donor specific anti-HLA antibodies detected by Luminex Single Antigen/specificity bead assay including weakly reactive antibodies that would not be detected by a flow cross match
2. Intolerance to any drug that will be used as part of the IS regimen.
3. Poorly controlled diabetes with an A1C of >8%.
4. Blood Pressure (BP): systolic blood pressure (SBP) > 140mmHg or DBP >90 mmHg despite treatment with antihypertensive agents. If the BP is greater than 140/90 chart review and discussion with the patient will be done to establish that BP is in good control.
5. Other exclusion criteria including significant renal or hepatic dysfunction
6. For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
7. Active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Quantiferon gold assay will be used to determine TB infection.
8. Invasive aspergillus, histoplasmosis, and coccidioidomycosis infection or other opportunistic infection within 1 year prior to study entry.
9. Current malignancy or treated malignancy with estimated recurrence rate >50% at 5 years, except for completely resected squamous or basal cell carcinoma of the skin
10. Known active alcohol or substance abuse.
11. Active infections (except mild skin and nail fungal infections).
12. Active peptic ulcer disease or gastritis, symptomatic gallstones, or portal hypertension.
13. Use of any investigational agents within 4 weeks of screening or 5 half-lives of the investigational product/ medication, whichever is longer. Investigational products with prolonged invivo effects will require a wash-out period that aligns with the biochemical and physiologic effects of the agent prior to the initiation of this protocol. If the half life of the experimental agent is not known, participation in the study will be addressed with the study team and documented in the study record.
14. Any investigational agents/products that could potentially interfere with the safety and/or efficacy of the procedure being studied will be addressed with the study team and documented in the study record.
15. Administration of live attenuated vaccine(s) within 2 months of enrollment.
16. Any medical condition that, in the opinion of the investigator, will interfere with safe study completion.
17. Positive screen for polyoma (BK) viremia at time of screening.
18. CKD stage 4 or 5
19. Severe co-existing cardiac disease, characterized by any one of these conditions:

    1. Recent myocardiol infarction (MI) (within 1 year)
    2. Evidence of ischemia on functional cardiac exam within the last year. These include persantine thallium stress test and/or coronary angiogram which will be performed in any patient with a history of an MI
    3. Left ventricular ejection fraction < 45%
    4. Valvular disease requiring replacement with prosthetic valve
20. Substance use that in the opinion of the investigator would interfere with compliance with the study requirements.
21. Past or current medical problems or findings from medical history, physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Levels of intact PTH | From baseline to week 52 (year 1)
  The primary efficacy endpoint is attainment of levels of intact PTH that are in the normal target range and at least a doubling of the baseline intact PTH level prior to transplantation
Incidence of Adverse Events | From baseline to Year 1
  The primary safety endpoint is the incidence of adverse events related to the transplant procedure or immunosuppression, incidence of post- transplant infections and malignancies, incidence of de novo sensitization

SECONDARY OUTCOMES:
Dose of oral calcium supplements and calcitrol | From baseline to week 52 (year 1)
  50% reduction from baseline in the oral dose of calcium supplements and in the oral dose of calcitriol with maintenance of stable serum calcium in normal range in patients taking conventional therapy with calcium salts and calcitriol
Dose of subcutaneous parathyroid hormone (PTH) replacement therapy | From baseline to week 52 (year 1)
  Reduction by 50% or greater in the dose of subcutaneous PTH replacement therapy with maintenance of serum calcium in the normal target range
PTH replacement therapy | From baseline to week 52 (year 1)
  Discontinuation of PTH replacement therapy with maintenance of serum calcium in the normal target range while taking 1000 mg or less of elemental calcium in the form of calcium supplements.

OTHER OUTCOMES:
Quality of Life measurement | From baseline to Year 1
  An exploratory endpoint is an improvement in one or more quality of life measurements comparing baseline and 3 months post-transplant using the Short Form 36 (SF36) survey and the Hypoparathyroidism Experience Scale (HPES)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stock, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, informed consent, clinical study report, and de-identified individual participant data (IPD) collected in this trial will be made available to other researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon completion of the clinical study report and publication of the trial outcomes.
Access Criteria: Researchers may contact Dr. Peter Stock, MD, PhD at UCSF by contacting the primary contact listed in this CT.GOV record.